CLINICAL TRIAL: NCT02319187
Title: Irinotecan Plus S1 Versus S1 in Patients With Previously Treated Advanced Esophageal Squamous Cell Carcinoma (ESWN 01 Trial): a Phase 3, Prospective,Multicenter, Randomised Study
Brief Title: Irinotecan Plus S1 Versus S1 in Patients With Previously Treated Advanced Esophageal Cancer: ESWN 01 Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jing Huang, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-064
Record Dates: First submitted 2014-12-09; First posted 2014-12-18 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-04

CONDITIONS: Esophageal Neoplasms
Keywords: Esophageal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms | interventions — S 1 (combination); Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): S1
  Interventions: Drug: S1
- Arm B (Experimental): S1 and irinotecan
  Interventions: Drug: S-1; Drug: irinotecan

INTERVENTIONS:
Drug: S1 — S1 80mg to 120 mg per day on Days 1-14, every 21 days
  Arms: Arm A
Drug: S-1 — S1 80mg to 120 mg per day on Days 1-10, every 14 days;
  Arms: Arm B
Drug: irinotecan — irinotecan 160mg/m2 d1, every 14 days
  Arms: Arm B

SUMMARY:
Esophageal cancer is a highly aggressive malignancy with a poor overall outcome.

The purpose of this study is to evaluate the progression free survival and safety of irinotecan plus S1 versus S1 alone in the patients with previously treated advanced esophageal cancer

DETAILED DESCRIPTION:
Two arms, phase 3 study of irinotecan plus S1 versus S1 alone in previously treated patients with recurrent or metastatic esophageal cancer. 240 Patients will be enrolled in this trial. The primary objective of this study is to determine the PFS of the two arms. One arm is as follows: irinotecan 160 mg/m2 will be administered as an intravenous infusion over 60 minutes on Days 1, followed by S1 80mg to 120 mg per day on Days 1-10, every 14 days per cycle. The other arm is S1 80mg to 120 mg per day on Days 1-14, every 21 days per cycle.This study will also include the investigation of UGT1A1polymorphisms in the study population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven esophageal squamous cell carcinoma;
* 18 ≤ age ≤ 70;
* ECOG 0-2;
* Previously Treated with platinum or paclitaxel based regimen;
* Uni-dimensionally measurable disease (CT or MRI as per RECIST);
* Patients should have a projected life expectancy of at least 3 months;
* Completion of baseline quality of life questionnaire
* Adequate bone marrow functions (ANC ≥ 1,500/ul, blood platelet ≥ 100,000/ul, haemoglobin ≥ 10g/dl);
* Adequate renal functions(serum creatinine ≤ 1.5mg/dl)
* liver functions (serum bilirubin ≤ 1.5UNL, AST/ALT ≤ 3 times(normal value)
* Written informed consent

Exclusion Criteria:

* Previous chemotherapy with 5-FU or irinotecan after recurrence or metastasis;
* adjuvant chemotherapy with 5-FU-based chemotherapy within 6 months prior to the start of study treatment;
* Active infection requiring antibiotics
* Pregnant, lactating women
* Psychiatric illness, epileptic disorders
* Concurrent systemic illness not appropriate for chemotherapy
* History of other malignancy within 5 years except for non-melanoma skin cancer, cervix in situ carcinoma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 2

SECONDARY OUTCOMES:
Adverse Events | 2 year
overall survival | 3 year
response rate | 1.5 year
quality of life | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, M.D., Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Jing Huang, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (13):
- China (13):
  - Hebei four Hospital, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Xinxiang Medical College, Xinxiang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Wuhan, Hubei
  - Mongolia Chifeng Hospital, Chifeng, Inner Mongolia
  - Ordos Central Hospital, Ordos, Inner Mongolia
  - Jiangsu Taizhou peoples Hospital, Taizhou, Jiangsu
  - Qinghai Cancer Hosptal, Xining, Qinghai
  - Shanxi Province Cancer Hospital, Taiyuan, Shanxi
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing
  - Hunan Cancer Hospital,the Affiliated Cancer Hospital of Xianya School of Medicine, Changsha
  - Herbin Medical University Cancer Hospital, Herbin
  - Henan Cancer Hospital, Zhengzhou

REFERENCES:
- [Derived] Huang J, Xu B, Liu Y, Huang J, Lu P, Ba Y, Wu L, Bai Y, Zhang S, Feng J, Cheng Y, Li J, Wen L, Yuan X, Ma C, Hu C, Fan Q, Wang X. Irinotecan plus S-1 versus S-1 in patients with previously treated recurrent or metastatic esophageal cancer (ESWN 01): a prospective randomized, multicenter, open-labeled phase 3 trial. Cancer Commun (Lond). 2019 Apr 2;39(1):16. doi: 10.1186/s40880-019-0359-7. PMID 30940189